CLINICAL TRIAL: NCT05643092
Title: Biomarker and Imaging Package Study in Immune Effector Cell-Associated Neurotoxicity Syndrome
Status: Recruiting | Type: Observational
Sponsor: zhang shoulong (Other)
Collaborators: Jinan Military General Hospital (Other); Changhai Hospital (Other)
Responsible Party: Sponsor-Investigator, zhang shoulong, Principal Investigator, Hebei Medical University
Organization: Hebei Medical University (Other)
Other Study IDs: 168
Record Dates: First submitted 2022-11-21; First posted 2022-12-08 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Immune Effector Cell Associated Neurotoxicity Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
CAR T-cell therapy is a promising innovative therapy for hematological malignancies. Immune effectors cells-associated neurotoxicity syndrome (ICANS) is a significant complication of CAR therapy. The goal of this study is to understand what brain mechanisms become disrupted when patients experience ICANS. The study will test the hypothesis that cerebrospinal fluid catecholamines and multimodal magnetic resonance imaging are affected in this disorder.

To test this hypothesis, the study will measure cerebrospinal fluid catecholamines in ICANS patients and evaluate brain magnetic resonance imaging for these participants. This study may contribute to knowledge about brain biomarkers and imaging of ICANS, which will greatly aid in ICANS detection and prevention.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be ≥ 18 years of age at signing of informed consent.
* Subjects are scheduled to receive CAR T-cell treatment.

Exclusion Criteria:

* Refusal to sign the informed consent
* Subjects having previously been treated with CAR-T therapy.
* Subjects with clinically significant active bleeding, history of intracranial bleeding, or is at risk for intracranial bleeding
* Subjects presenting primary CNS lymphoma
* Pacemaker or other implanted electrical device incompatible with the MR environment
* Subjects with a neurodegenerative disease (PD, AD)
* Subjects with a previous or evolving neurological pathology
* Pregnant or breastfeeding women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective observational study using a consecutive patient sample.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of CAR-T-associated Neurotoxicity | up to 3 years post CAR T-cell infusion
  The incidence of CAR-T-associated neurotoxicity of any grade defined by ASTCT

SECONDARY OUTCOMES:
To identify biomarkers for ICANS | up to 1 years post CAR T-cell infusion
  Serum and cerebrospinal fluid cytokines, neurocognitive assessments (Montreal Cognitive Assessment)
MRI scans for ICANS | up to 1 years post CAR T-cell infusion
  Lesion location associated with severity of ICANS

CONTACTS AND LOCATIONS:
Overall Officials: Shoulong Zhang, Principal Investigator — 980th Hospital
Locations (1):
- 980th Hospital, Shijiazhuang, Hebei, China